CLINICAL TRIAL: NCT06621368
Title: Effect of Two Years of Resistance Training on Muscular Strength, Body Composition, Functional Fitness, Metabolic Biomarkers, Cognition, and Cardiac Parameters in Postmenopausal Women: Longitudinal Study Active Aging
Brief Title: Effect of Two Years of Resistance Training on Health Status in Postmenopausal Women: Longitudinal Study Active Aging.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Edilson Serpeloni Cyrino, Principal investigator, PhD, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GEPEMENE 2024b
Record Dates: First submitted 2024-09-12; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Aging
Keywords: bone mineral density; health´s women; skeletal muscle mass; motor performance; strength training; metabolism
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group = participants maintained their usual activities normally (No Intervention): Participants maintained their ususal activities normally
- exercise group = participants performed two years of strength training (Experimental): Participants will performed two years of strength training
  Interventions: Other: Exercise; Other: Control-no treatment

INTERVENTIONS:
Other: Exercise — the RT program will consist of eight exercises for different body segments, namely: vertical bench press, horizontal leg press, low row, leg extension, scott curl, leg curl, triceps pulley and seated calf raise. Every 12 weeks of training, the program will be restructured with changes in the order in which the exercises are performed, the number of sets, the number of repetitions or the training system in an attempt to avoid a supposed adaptive plateau. The protocols in each stage will follow the recommendations for prescribing RT for the elderly, aiming at improving strength and hypertrophy, namely: a combination of single-joint and multi-joint exercises (free weights and machines), slow or moderate execution speed (ratio 1:2 for concentric and eccentric muscle actions, respectively), one to three sets of multiple repetitions, 8-12 RM or 10-15 RM, with recovery intervals between sets of one to two minutes, and a training frequency of two to three weekly sessions, on alternate days.
  Other Names: Resistance traning
  Arms: exercise group = participants performed two years of strength training
Other: Control-no treatment — Participants will maintain their daily activities.
  Arms: exercise group = participants performed two years of strength training

SUMMARY:
Aging is a natural process of the life cycle that can result in morphological, neuromuscular, metabolic, physiological, cognitive and behavioral changes that can compromise quality of life, autonomy, self-esteem, health and life expectancy, especially in the elderly. On the other hand, resistance training (RT) has been widely recommended for the elderly population, due to the numerous health benefits it brings, such as increased strength and muscle mass, reduced body fat, increased bone mineral content and density, and improved cardiometabolic profile, among others. However, the effectiveness of RT in attenuating or reversing the deleterious effects of aging has been analyzed by studies conducted, in most cases, over relatively short periods, i.e., eight to 24 weeks. Considering that recent investigations have demonstrated a wide variation in the adaptive responses to RT in this population, it is likely that many of these responses are time-dependent. Additionally, the influence of important mediators and moderators in this process, especially training intensity and volume, dietary habits, the presence or absence of diseases and degenerative processes that cause disability, and the use of polypharmaceuticals, has not yet been well established. Therefore, based on the Active Aging Longitudinal Study, a research project initiated in 2012, it is intend to analyze whether or not RT practice can produce positive and lasting adaptive responses on muscle strength, body composition, functional fitness, cognition, cardiometabolic biomarkers, and cardiac function in postmenopausal women, based on a randomized controlled clinical trial over a long period of time (two years). In addition, mediation and moderation analyses will be used to understand the real impact of RT on the outcomes to be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older;
* physically independent;
* not have cardiovascular, musculoskeletal or metabolic limitations that prevent the practice of physical exercises or the execution of motor tests;
* not being on hormone replacement therapy;
* not being involved in physical exercise more than once a week, over the six months prior to the start of the study.

Exclusion Criteria:

* not participating in at least 85% of the training and not attending the assessments.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-11-23 (Estimated)

PRIMARY OUTCOMES:
Body Fat | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  Dual-energy x-ray absorptiometry examinations were performed in a Lunar Prodigy device, model NRL 41990 (General Electric, Madison, WI), to determine the total, regional lean soft tissue (LST), appendicular LST (ALST), and the total body, trunk, gynoid, and android fat masses (all these outcomes are presented in kilograms). Participants were instructed to remove all metal objects before scanning to minimize possible estimation errors. Scans were performed with participants lying in the supine position along the table's longitudinal centerline axis. Feet were secured together at the toes to immobilize the legs while the hands were maintained in a pronated position within the scanning region. A skilled researcher carried out both calibration and analysis, following the manufacturer's recommendations. The software generated standard lines that separated the limbs from the trunk and head.
Muscle mass | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  Dual-energy x-ray absorptiometry examinations were performed in a Lunar Prodigy device, model NRL 41990 (General Electric, Madison, WI), to determine the total, regional lean soft tissue (LST), appendicular LST (ALST), and the total body, trunk, gynoid, and android fat masses (all these outcomes are presented in kilograms). Participants were instructed to remove all metal objects before scanning to minimize possible estimation errors. Scans were performed with participants lying in the supine position along the table's longitudinal centerline axis. Feet were secured together at the toes to immobilize the legs while the hands were maintained in a pronated position within the scanning region. A skilled researcher carried out both calibration and analysis, following the manufacturer's recommendations. The software generated standard lines that separated the limbs from the trunk and head.

SECONDARY OUTCOMES:
Cardiovascular risk factors | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  HDL-c (mg/dL), LDL-c (mg/dL), Total cholesterol (mg/dL), Glucose (mg/dL), triglycerides(mg/dL), C-reactive protein (mg/dL)
Cardiac function | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  Echocardiography exams were performed accord- ing to current guidelines [18], at baseline and the end of the investigation, by an experienced echocardi- ographer blinded to patient status and group assign- ment, using a Philips ultrasound machine, model iE33 (Philips Medical Solutions, Noord Brabant, The Netherlands), equipped with an S5-1 and X5-1 transducer. According to current recommendations, cardiac chamber dimensions, volumes, and left ven- tricular mass were measured. Mitral inflow velocities were assessed using a pulsed-wave Doppler in the apical four-chamber view, with the sample volume placed between the tips of the mitral leaflets; veloci- ties were recorded at end-expiration. Tissue Doppler velocities were acquired at end-expiration, in the api- cal four-chamber view, with the sample positioned at the septal and lateral mitral annulus for determination of systolic (S'), early diastolic (E'), and late diastolic (A') velocities.
MoCA | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  The Brazilian version ofthe Montreal Cognitive Assessment (MoCA) was used to analyze the global cognitive function. The MoCA is a screening tool composed of 12 individually punctuated tasks grouped into eight cognitive domains. The total score ranges from 0 to 30 (higher values reflect better cognition). Cognitive domains and their respective punctuations are as follows: short-term memory (delayed recall, 5 points); visuospatial abilities (cube drawing, 1 point, clock drawing, 3 points); executive function (trail making test, 1 point; phonemic verbal fluency, 1 point; verbal abstraction, 2 points); attention, concentration, andwork- ing memory (cancelation, 1 point; subtraction, 3 points; digit span, 2 points); language (naming, 3 points; sentence repetition, 2 points); and orientation to time (3 points) and space (3 points).
Stroop test | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  The Stroop test version used in the present study consisted of 36 tasks. In every trial, one cue appeared at the top part of the screen and the bottom two response options, one matched and one mismatched. Participants had to press the directional button (< or >) corresponding to the position ofthe correct response as quickly and accurately as possible. The test consisted of three stages with 12 trials each: (I-congruent) an inked rect- angle (green, black, red, or blue) appeared, and participants had to choose the response corresponding to the ink name; (II- neutral) a color name (green, black, red, or blue) appeared in white ink, and participants had to choose the option corresponding to the color name; (III-incongruent) a color name appeared at the top of the screen in a different ink color (e.g., the word black in green ink). The participants had to respond to the ink color, not the color name (e.g., green in this example).
Set shifting | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  The Trail Making Tests parts A and B were used to assess set shifting. Part A assesses the psychomotor speed and requires the participant to draw lines that connect encircled numbers sequentially, such as drawing a line from 1 to 2, 2 to 3, 3 to 4, and so on. Part B consists ofencircled numbers and letters. Participants were instructed to draw a line as quickly and as accurately as possible from 1 to A, A to 2, 2 to B, B to 3, and so on, until they completed the task. We recorded the time (in seconds) they took to complete each task. We calculated the difference between part B and part A completion times to index set shifting. Smaller difference scores indicate better set shifting.
Verbal fluency tasks | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  Participants were asked to say asmany words as possible within 60 s (31). In the first trial, par- ticipants had to produce words starting with the letter "F" (letter fluency) and produce the name of animals (category fluency). The final score refers to the number ofwords correctly spoken in 60 s.
Depressive symptoms | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  The 15-item Geriatric Depres- sion Scale (GDS-15): The GDS-15 comprises 15 dichotomic items (yes or not) concerning different characteristics of geriatric depression as cognitive decline and somatic symptoms, with the final score ranging from 0 to 15, where the higher scores are worse.
Anxiety symptoms | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  Beck Anxiety Inventory (BAI): The BAI comprises 21 items (statements) about different anxiety symptoms with a 4-point Likert scale, with the final score ranging from 0 to 63, where the higher scores are worse.
Bone | from begining (November 2023) to the end 48 weeks of resistance training (November 2026)
  Dual-energy x-ray absorptiometry examinations were performed in a Lunar Prodigy device, model NRL 41990 (General Electric, Madison, WI), to determine the total and regional bone mineral density (cm/m²). Participants were instructed to remove all metal objects before scanning to minimize possible estimation errors. Scans were performed with participants lying in the supine position along the table's longitudinal centerline axis. Feet were secured together at the toes to immobilize the legs while the hands were maintained in a pronated position within the scanning region. A skilled researcher carried out both calibration and analysis, following the manufacturer's recommendations. The software generated standard lines that separated the limbs from the trunk and head.

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nabuco HCG, Tomeleri CM, Sugihara Junior P, Fernandes RR, Cavalcante EF, Antunes M, Ribeiro AS, Teixeira DC, Silva AM, Sardinha LB, Cyrino ES. Effects of Whey Protein Supplementation Pre- or Post-Resistance Training on Muscle Mass, Muscular Strength, and Functional Capacity in Pre-Conditioned Older Women: A Randomized Clinical Trial. Nutrients. 2018 May 3;10(5):563. doi: 10.3390/nu10050563. PMID 29751507
- [Background] Dos Santos L, Cyrino ES, Antunes M, Santos DA, Sardinha LB. Sarcopenia and physical independence in older adults: the independent and synergic role of muscle mass and muscle function. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):245-250. doi: 10.1002/jcsm.12160. Epub 2016 Nov 8. PMID 27897417